CLINICAL TRIAL: NCT05119452
Title: Screening for Flare After Discontinuation of Biological/Targeted Synthetic Disease Modifying Anti-rheumatic Drug (b/tsDMARD) in Rheumatoid Arthritis
Brief Title: Screening for Flare After b/tsDMARD Discontinuation in Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Medical University of Graz (Other); Medical University Innsbruck (Other); Hospital Hietzing (Other); Krankenhaus Bruneck (Other)
Responsible Party: Principal Investigator, Dr. Peter Mandl, Ap. Prof. Priv.-Doz. Dr. Peter Mandl, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1389/2020
Record Dates: First submitted 2021-11-02; First posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab; golimumab; Certolizumab Pegol; tocilizumab; sarilumab; Etanercept; Interleukin 1 Receptor Antagonist Protein; GLPG0634; tofacitinib; baricitinib

STUDY DESIGN:
Intervention Model Description: At baseline, patients will be randomised in a 1:1 ratio in an "Assisted monitoring" (arm A) or a "Clinical monitoring" (arm B) arm respectively.
Who Masked: Participant, Investigator
Masking Description: After checking the inclusion- and exclusion criteria and after the patients´ consent the study investigator contacts the administrative office of the coordinating center. The online computerised randomisation algorithm "Randomizer for Clinical Trials by the Medical University of Vienna (MUW) will be used for randomisation for all centres.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assisted monitoring (Other): In the Assisted monitoring arm, C-reactive protein and musculoskeletal ultrasound information will be made available to the clinical assessors who, at each time-point will use this information, along with information from the clinical examination, to identify patients experiencing recurrence of inflammation which will then be counted as subclinical flare according to predefined criteria.
  Interventions: Other: Discontinuation of biological/targeted synthetic disease modifying anti-rheumatic drug (b/tsDMARD)
- Clinical monitoring (Other): In the Clinical monitoring arm, the results of C-reactive protein and musculoskeletal ultrasound information will be recorded but will not be made available to the clinical assessor who at each time-point will make the decision on whether the patient is experiencing or has experienced a clinical flare according to predefined criteria based on information from the clinical examination.
  Interventions: Other: Discontinuation of biological/targeted synthetic disease modifying anti-rheumatic drug (b/tsDMARD)

INTERVENTIONS:
Other: Discontinuation of biological/targeted synthetic disease modifying anti-rheumatic drug (b/tsDMARD) — The biological/targeted synthetic disease modifying anti-rheumatic drug will be discontinued in both arms at baseline
  Other Names: b/tsDMARD: Adalimumab, Infliximab, Golimumab, Certolizumab pegol, Tocilizumab, Sarilumab, Etanercept, Anakinra, Filgotinib, Updacitinib, Tofacitinib, Baricitinib

SUMMARY:
To evaluate whether stringent follow-up consisting of combined laboratory and ultrasound surveillance is superior to clinical monitoring alone to maintain clinical remission in rheumatoid arthritis.

DETAILED DESCRIPTION:
Randomized, controlled, parallel-group, multi-centre study in which patients with rheumatoid arthritis treated with biological/targeted synthetic disease modifying antirheumatic drug (b/tsDMARD) in mono- or combination therapy with conventional synthetic disease modifying antirheumatic drug (csDMARD) in a stable dosage and interval for ≥6 months with low disease activity or remission will receive an power Doppler musculoskeletal ultrasound examination (PDUS) and monitoring of C-reactive protein (CRP) levels at baseline and several timepoints within a 24 month study period (primary endpoint) and within a 48 month long-term extension. At baseline, b/tsDMARD medication will be withdrawn in all patients, who will be randomized in a 1:1 ratio in an "Assisted monitoring" (arm A) or a "Clinical monitoring" (arm B) arm respectively. Further stratification for remission vs. low disease activity and mono- vs combination therapy will be implemented in the randomisation process. In arm A, CRP and PDUS information will be made available to the clinical assessors who, at each time-point will use this information along with that from clinical examination, to identify patients experiencing recurrence of inflammation which will then be counted as subclinical flare according to predefined criteria. In arm B the results of CRP and PDUS will be recorded but will not be made available to the clinical assessor who will have to identify clinical flares according to predefined criteria based on information from the clinical examination only.

ELIGIBILITY:
Inclusion Criteria:

Patients with rheumatoid arthritis classified by the American College of Rheumatology/European League Against Rheumatism classification criteria

* biological disease-modifying anti-rheumatic drug (bDMARD) or targeted synthetic disease-modifying anti-rheumatic drug (tsDMARD) treatment in monotherapy or in combination therapy with conventional synthetic disease-modifying anti-rheumatic drug (csDMARD) in a stable dosage and interval for ≥6 months. Previous extension of bDMARD or tsDMARD interval will also be accepted. bDMARDs and tsDMARDs will include all currently available originator and biosimilar compounds, with the exception of rituximab and its biosimilar compounds
* No swollen joint by 28-joint count at baseline, and screening
* C-reactive protein of ≤0.5mg/dL at baseline AND history of C-reactive protein >0,5mg/dl related to rheumatoid arthritis activity
* Clinical disease activity index ≤10
* Shared decision between patient and physician to attempt b/tsDMARD withdrawal
* Willing and able to understand and follow the study procedures
* Written informed consent
* Female and male subjects aged ≥ 18 years

Exclusion Criteria:

* History of or current extra-articular manifestation of rheumatoid arthritis, with exception of rheumatoid nodules
* Systemic glucocorticoid treatment in the past 3 months
* Intraarticular injection with glucocorticoids in the past 1 month
* Joint replacement surgery other than total knee or hip arthroplasty or complete joint destruction
* Power Doppler signal ≥2 in any assessed joint and/or tendon at screening or baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects without a clinical flare until week 24 | week 24
  Proportion of subjects without a clinical flare

SECONDARY OUTCOMES:
Proportion of subjects without a clinical flare | week 48
  Proportion of subjects without a clinical flare
Time to clinical flare (days) | study period
  Time to clinical flare (days)
28 swollen joint count | week 24
  28 swollen joint count, scale 0 (best) - 28 (worse)
28 tender joint count | week 24
  28 tender joint count, scale 0 (best) - 28 (worse)
Proportion of subjects with a clinical flare in the assisted monitoring arm vs. clinical monitoring arm, the latter stratified according to b/tsDMARD reinitiation | week 24
  Proportion of subjects with a clinical flare in the assisted monitoring arm vs. clinical monitoring arm, the latter stratified according to b/tsDMARD reinitiation
Proportion of patients in low disease activity or remission based on simplified disease activity index | week 24
  Proportion of patients in low disease activity or remission based on simplified disease activity index
Proportion of patients in low disease activity or remission based on simplified disease activity index | week 48
  Proportion of patients in low disease activity or remission based on simplified disease activity index
Patient's global assessment | week 24
  Patient's global assessment, scale 0 (best) - 100 (worst)
Evaluator's global assessment | week 24
  Evaluator's global assessment, scale 0 (best) - 100 (worst)
C-reactive protein | week 24
  C-reactive protein, scale 0 (best) - infinite (worst)
Radiographic progression | at week 48 weeks from baseline
  change in Sharp Van der Heijde score, scale 0 (best) - 488 (worse)
Health Assessment Questionnaire Disability Index | week 24
  Health Assessment Questionnaire Disability Index, scale 0 (best) - 3.0 (worse)
World Health Organization Quality of Life Questionnaire | week 24
  World Health Organization Quality of Life Questionnaire, scale 0 (worse) - 100 (best)
Morning stiffness | week 24
  Morning joint stiffness, (minutes), scale 0 (best) - infinite (worst)
Fatigue | week 24
  Fatigue, visual analogue scale, scale 0 (worse) - 100 (best)